CLINICAL TRIAL: NCT05704855
Title: A Remotely-Delivered, Combined Exercise Training Program for Cognitive Function in Women Living With and Beyond Breast Cancer: A Feasibility Study
Brief Title: A Combined Exercise Training Program for Women Living With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Linda Trinh, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BCSPilot01
Record Dates: First submitted 2023-01-10; First posted 2023-01-30 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: physical activity; chemotherapy treatment; cancer-related cognitive impairment; feasibility; mental health
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Psychological Well-Being | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two conditions: combined exercise (aerobic + resistance training) or stretching/toning (active control). They will receive a home-based program lasting 1 hour on 3 days per week for 12 weeks. Randomization will be performed using a computer-generated program in blocks of four for even distribution between study conditions. BCS will be assigned in a 1:1 ratio to one of two study conditions, stratified by treatment type (anthracycline vs. non-anthracycline chemotherapy; hormonal vs. no hormonal therapy).
Who Masked: Participant
Masking Description: The participants will only be aware that the researchers are comparing two exercise conditions and therefore will be blinded to the study hypotheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Exercise + Behavioural Counselling (Experimental): The combine exercise intervention will consist of three 30-minute, supervised, remotely-delivered resistance training classes as well as three 30-minute, unsupervised aerobic training (i.e., walking) items each week. Participants will also participate in bi-weekly, 30-40 minute, remotely-delivered behavioural counselling sessions delivered via videoconferencing (i.e., Zoom). The program will be taught by a Registered Kinesiologist via videoconferencing (i.e., Zoom). Participants will be asked to participate in the intervention for 8 weeks.
  Interventions: Behavioral: Combined Exercise + Behavioural Counselling
- Active Control (Active Comparator): The active control group will participate in three 30-minute, supervised, remotely-delivered classes targeting balance and flexibility. The program will be delivered at a low-intensity by a Registered Kinesiologist via videoconferencing (i.e., Zoom). Participants will be asked to participate in the program for 8 weeks.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Combined Exercise + Behavioural Counselling — The combine exercise intervention will consist of three 30-minute, supervised, remotely-delivered resistance training classes as well as three 30-minute, unsupervised aerobic training (i.e., walking) sessions each week. Participants will also participate in bi-weekly, 45-60 minute, remotely-delivered, group-based behavioural counselling sessions delivered via videoconferencing (i.e., Zoom). Participants will be asked to participate in the intervention for 8 weeks.
  Arms: Combined Exercise + Behavioural Counselling
Behavioral: Active Control — The active control group will participate in three 30-minute, supervised, remotely-delivered classes targeting balance and flexibility. The program will be delivered at a low-intensity by a Registered Kinesiologist via videoconferencing (i.e., Zoom). Participants will be asked to participate in the program for 8 weeks.
  Arms: Active Control

SUMMARY:
Women living with and beyond breast cancer are at a heightened risk for experiencing adverse mental health outcomes and declines in cognitive function following chemotherapy treatment. Women living with and beyond breast cancer have reported increased levels of anxiety and depression during the COVID-19 pandemic which may have significantly impacted their quality of life (QoL). Physical activity (PA) may be used to manage mental health and improve cognitive function in women living with and beyond breast cancer. Research is needed to assess the feasibility of a supervised, remotely delivered, combined (i.e., aerobic + resistance) exercise program to improve cognitive function and manage adverse mental health in women living with and beyond breast cancer. This study will pilot an 8-week, remotely delivered, combined (i.e., aerobic + resistance) exercise and behavioural counselling intervention on cognitive function and mental health outcomes (i.e.,anxiety, depression, self-efficacy and self esteem) in women living with breast cancer who received chemotherapy treatment within 12-48 months.

DETAILED DESCRIPTION:
Women living with and beyond breast cancer who received chemotherapy treatment are at a heightened risk for experiencing adverse mental health outcomes (i.e., anxiety, depression, self-efficacy and self esteem) and declines in cognitive function (i.e., impairments to memory, learning, concentration, reasoning, executive function, attention, processing speed and/or visual-spatial skills deficits) compared to those without a history of cancer. These effects may be worsened among those who received chemotherapy treatment and may persist for up to 5 and 20 years following chemotherapy treatment completion, respectively. The COVID-19 pandemic has exacerbated existing adversities in the mental health of women living with and beyond breast cancer due to reduced social opportunities, greater sedentary time, fear of susceptibility to the virus and barriers to in-person support services. Physical activity (PA) may be used to manage mental health adversities and improve QoL among women living with and beyond breast cancer. In addition, preliminary evidence has demonstrated the potential mediating effect of PA on cognitive impairments among women living with and beyond breast cancer. Remote-based interventions could be an effective option to increase PA during the COVID-19 pandemic while maintaining physical distancing protocols. In addition, the combination of exercise with group-based counselling has been found to be feasible and provide favourable improvements in depression, self-efficacy, social support, and quality of life and long-term PA maintenance among women living with and beyond breast cancer, compared to exercise interventions alone. However, no studies have evaluated the feasibility and impact of a supervised, remotely delivered, combined (i.e., aerobic and resistance) exercise + behaviour counselling program on mental health and cognitive function in women living with and beyond breast cancer following chemotherapy treatment. Using a mixed-method approach, this study will address these gaps by evaluating the feasibility of a supervised, remotely delivered combined (i.e., aerobic and resistance) exercise and behavioural counselling program for mental health and cognitive function in women living with and beyond breast cancer. This project is necessary given the remote-based format of exercise delivery that has been adopted because of the COVID-19 pandemic and the need for programs to be adapted to an environment that is safe and reliable to deliver to women living with and beyond breast cancer.

ELIGIBILITY:
* 40 - 65 years of age
* primary diagnosis of stage I-III breast cancer (non-metastatic)
* received chemotherapy within the past 12-48 months from enrollment
* experience mild cognitive impairment as determined by the TICS [scores between 28-31 to separate individuals with dementia (range a to b) and normal cognition (range c to d)] (Knopman et al., 2010)
* self-reported low-active defined as <3 days of exercise (<20 min/day) per week in the previous six months (Godin & Shephard, 1985)
* physician clearance to participate in testing and exercise
* no previous invasive cancer
* no neurological or musculoskeletal co-morbidity inhibiting exercise
* access to a webcam and internet for videoconferencing
* English fluency.

Exclusion Criteria:

* previous invasive cancer
* neurological or musculoskeletal co-morbidity inhibiting exercise

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Enrolment rate | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Participant enrolment rate will be one measure of feasibility. This will be calculated by measuring the amount of participants who enrolled in the intervention, divided by the number of participants who were assessed for eligibility.
Adherence rate | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Adherence rate of participants to the intervention, will be one measure of feasibility. This will be measured by calculating the number of exercise sessions participants attend, divided by the total number of exercise sessions that took place in the intervention.
Attrition rate | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Attrition will be one measure of feasibility. This will be measured by calculating the number of participants who did not complete the intervention, divided by the number of participants who completed the entirety of the intervention
Burden and satisfaction | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Burden and satisfaction scores will be one measure of feasibility. This will be assessed using a researcher-generated 15-item questionnaire that asks participants about their experience with the intervention and assessments. Participants will rate items using a 5-point Likert scale (1= 'strongly disagree', 5 = 'strongly agree').
Adverse events | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Adverse events will be one measure of feasibility. This will be assessed as an unexpected and severe medical problem or injury that occurs during the exercise classes.

SECONDARY OUTCOMES:
Executive/Attention | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Flanker Inhibitory Control and Attention Test tests the ability to inhibit visual attention to irrelevant task dimensions. A scoring algorithm integrates accuracy and reaction time yielding scores from 0 to 10. There are 40 trials and the average time to complete the task is 4 minutes.To interpret individual performance, one can evaluate all three types of scale scores in which higher scores indicate higher levels of ability to attend to relevant stimuli and inhibit attention from irrelevant stimuli.
Episodic Memory | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Picture Sequence Memory Test involves a presentation of stimuli which are pictured objects and activities, thematically related but with no inherent order. For each trial, pictures appear in the center of the screen and then are moved 1 at a time into a fixed spatial order, as an audio file simultaneously describes the content of each. The score is based on the cumulative number of adjacent pairs of pictures remembered correctly over 3 learning trials. The test takes approximately 10 minutes. Higher scores indicate better episodic memory.
Language | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Picture Vocabulary Test involves single words that are presented via an audio file, paired simultaneously with 4 screen images of objects, actions, and/or depictions of concepts. The participant will pick the picture that matches the spoken word. Total administration time is approximately 5 minutes. To interpret individual performance, one can evaluate all three types of scale scores. A participant's age-adjusted scale score at or near 100 indicates vocabulary ability that is average for the age level. Scores around 115 suggest above-average vocabulary ability, while scores around 130 suggest superior ability - in the top 2 percent nationally for age, based on Toolbox normative data.
Crystallized Cognition | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). This composite includes the Picture Vocabulary and Reading Tests. This composite score is derived by averaging the normalized scores of each of the measures, and then deriving scale scores based on this 14 new distribution. An Age-Adjusted Scale Score, Fully Adjusted Scale Score, Unadjusted Scale Score and Age-Adjusted National Percentile are provided for the Crystallized Cognition Composite. Crystallized Cognition Composite is a more global assessment of individual and group verbal reasoning. Higher scores indicate higher levels of functioning.
Immediate Recall | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Auditory Verbal Learning Test (Rey) measures immediate recall. Unrelated words presented via audio recording and participant recalls as many as possible. he Rey is scored by taking the sum of the number of words recalled across all trials (possible range is 0-45 words). The raw score is most commonly used for interpretation of the Rey test, with higher scores reflecting better episodic memory.
Processing Speed | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Cognitive function will be assessed using the NIH toolbox cognition battery. The NIH toolbox cognition battery with computerized cognitive tasks and automated scoring was used (Weintraub et al., 2013). The Oral Symbol Digit Test measures speed of processing. Symbols on the screen are associated with a number, then presented with symbols without numbers. The Oral Symbol Digit Test is scored as the number of items answered correctly in 120 seconds (possible range is 0-144).Higher scores indicate better processing speed.
Self-reported anxiety and depression | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Measured using the Hospital Anxiety and Depression Scale (HADS), which is a 14-item questionnaire divided into two subscales of seven items each measuring anxiety (HADS-A) and depression (HADS-D). Two sub-scores (HADS-A and HADS-D) will be calculated with scores that vary from 0 to 21. Higher scores indicate more anxious/depressive symptoms (Zigmond & Snaith, 1983).
Self-efficacy | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Self-efficacy will be measured using the Breast Cancer Survivor Self Efficacy Scale. This is an 11-item Likert scale through which participants rate their responses from 1'strongly disagree' to 4, 'strongly agree'. A higher total score indicates better self efficacy.
Self-esteem | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Self-esteem will be measured pre-intervention and post-intervention (i.e., 8 weeks) using the Rosenberg Self-Esteem scale. This is a 10-item, likert style scale through which participants rate their responses from 1, 'strongly disagree' to 5, 'strongly agree'. Higher total scores indicate better self-esteem.
Objectively-assessed physical activity | Change from baseline (pre-intervention) to post-intervention (8 weeks).
  Objectively assessed PA was measured using Actigraph GTX3+ accelerometers (Pensacola, FL). Participants will wear the accelerometer on their non-dominant hip during waking hours for 7 consecutive days. Data will be downloaded in 60-s epochs and processed and converted to mean counts per minute in ActiLife software package (Version 6; Actigraph) to estimate daily minutes of light (101-1951 counts min-1), moderate (1952-5724 counts min-1), vigorous (≥ 5725 counts min-1), and total moderate-to-vigorous physical activity (MVPA; ≥ 1952 counts min-1) based on established cut-points (Freedson, Melanson, & Sirard, 1998). Estimated average daily minutes spent in each activity intensity category was calculated by dividing the number of minutes spent in each category by the total number of valid days worn.
Semi-structured qualitative interviews | Post-intervention (8 weeks).
  The researcher will conduct semi-structured qualitative interviews over videoconferencing that will ask participants about their experience with the study and intervention, including enjoyment, potential barriers faced, and how they felt mentally and cognitively during and after the intervention.
Therapeutic alliance | Post-intervention (8 weeks).
  Therapeutic alliance will be measured using the Working Alliance Inventory Short Revised (WAI-SR). This is a Likert scale through which participants rate their responses from 1, 'seldom', to 5, 'always'. A higher total score indicates better therapeutic alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Trinh, PhD, Principal Investigator — University of Toronto
Locations (1):
- Faculty of Kinesiology and Physical Education, University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Castellon SA, Ganz PA, Bower JE, Petersen L, Abraham L, Greendale GA. Neurocognitive performance in breast cancer survivors exposed to adjuvant chemotherapy and tamoxifen. J Clin Exp Neuropsychol. 2004 Oct;26(7):955-69. doi: 10.1080/13803390490510905. PMID 15742545
- [Background] Kesler SR, Kent JS, O'Hara R. Prefrontal cortex and executive function impairments in primary breast cancer. Arch Neurol. 2011 Nov;68(11):1447-53. doi: 10.1001/archneurol.2011.245. PMID 22084128
- [Background] Koppelmans V, Breteler MM, Boogerd W, Seynaeve C, Gundy C, Schagen SB. Neuropsychological performance in survivors of breast cancer more than 20 years after adjuvant chemotherapy. J Clin Oncol. 2012 Apr 1;30(10):1080-6. doi: 10.1200/JCO.2011.37.0189. Epub 2012 Feb 27. PMID 22370315
- [Background] Kesler S, Hadi Hosseini SM, Heckler C, Janelsins M, Palesh O, Mustian K, Morrow G. Cognitive training for improving executive function in chemotherapy-treated breast cancer survivors. Clin Breast Cancer. 2013 Aug;13(4):299-306. doi: 10.1016/j.clbc.2013.02.004. Epub 2013 May 4. PMID 23647804
- [Background] Argyriou AA, Assimakopoulos K, Iconomou G, Giannakopoulou F, Kalofonos HP. Either called "chemobrain" or "chemofog," the long-term chemotherapy-induced cognitive decline in cancer survivors is real. J Pain Symptom Manage. 2011 Jan;41(1):126-39. doi: 10.1016/j.jpainsymman.2010.04.021. Epub 2010 Sep 15. PMID 20832978
- [Background] Von Ah D, Tallman EF. Perceived cognitive function in breast cancer survivors: evaluating relationships with objective cognitive performance and other symptoms using the functional assessment of cancer therapy-cognitive function instrument. J Pain Symptom Manage. 2015 Apr;49(4):697-706. doi: 10.1016/j.jpainsymman.2014.08.012. Epub 2014 Sep 18. PMID 25240787
- [Background] Zimmer P, Baumann FT, Oberste M, Wright P, Garthe A, Schenk A, Elter T, Galvao DA, Bloch W, Hubner ST, Wolf F. Effects of Exercise Interventions and Physical Activity Behavior on Cancer Related Cognitive Impairments: A Systematic Review. Biomed Res Int. 2016;2016:1820954. doi: 10.1155/2016/1820954. Epub 2016 Apr 10. PMID 27144158
- [Background] Frank JS, Vance DE, Triebel KL, Meneses KM. Cognitive Deficits in Breast Cancer Survivors After Chemotherapy and Hormonal Therapy. J Neurosci Nurs. 2015 Dec;47(6):302-12. doi: 10.1097/JNN.0000000000000171. PMID 26447567
- [Background] Von Ah D, Habermann B, Carpenter JS, Schneider BL. Impact of perceived cognitive impairment in breast cancer survivors. Eur J Oncol Nurs. 2013 Apr;17(2):236-41. doi: 10.1016/j.ejon.2012.06.002. Epub 2012 Aug 14. PMID 22901546
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546
- [Background] Hartman SJ, Nelson SH, Myers E, Natarajan L, Sears DD, Palmer BW, Weiner LS, Parker BA, Patterson RE. Randomized controlled trial of increasing physical activity on objectively measured and self-reported cognitive functioning among breast cancer survivors: The memory & motion study. Cancer. 2018 Jan 1;124(1):192-202. doi: 10.1002/cncr.30987. Epub 2017 Sep 19. PMID 28926676
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] Weller IM, Thomas SG, Gledhill N, Paterson D, Quinney A. A study to validate the modified Canadian Aerobic Fitness Test. Can J Appl Physiol. 1995 Jun;20(2):211-21. doi: 10.1139/h95-015. PMID 7640647
- [Background] Champion VL, Ziner KW, Monahan PO, Stump TE, Cella D, Smith LG, Bell CJ, Von Ah D, Sledge GW. Development and psychometric testing of a breast cancer survivor self-efficacy scale. Oncol Nurs Forum. 2013 Nov;40(6):E403-10. doi: 10.1188/13.ONF.E403-E410. PMID 24161644
- [Background] Rosenberg M. Rosenberg self-esteem scale. Journal of Religion and Health. 1965 Jul.
- [Background] Hatcher RL, Gillaspy JA. Development and validation of a revised short version of the Working Alliance Inventory. Psychotherapy research. 2006 Jan 1;16(1):12-25.
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Carreira H, Williams R, Muller M, Harewood R, Stanway S, Bhaskaran K. Associations Between Breast Cancer Survivorship and Adverse Mental Health Outcomes: A Systematic Review. J Natl Cancer Inst. 2018 Dec 1;110(12):1311-1327. doi: 10.1093/jnci/djy177. PMID 30403799
- [Background] Jones JM, Saeed H, Katz MS, Lustberg MB, Forster VJ, Nekhlyudov L. Readdressing the Needs of Cancer Survivors During COVID-19: A Path Forward. J Natl Cancer Inst. 2021 Aug 2;113(8):955-961. doi: 10.1093/jnci/djaa200. PMID 33367655
- [Background] Aguinaga S, Ehlers DK, Cosman J, Severson J, Kramer AF, McAuley E. Effects of physical activity on psychological well-being outcomes in breast cancer survivors from prediagnosis to posttreatment survivorship. Psychooncology. 2018 Aug;27(8):1987-1994. doi: 10.1002/pon.4755. Epub 2018 Jun 1. PMID 29740914
- [Background] Aydin M, Kose E, Odabas I, Meric Bingul B, Demirci D, Aydin Z. The Effect of Exercise on Life Quality and Depression Levels of Breast Cancer Patients. Asian Pac J Cancer Prev. 2021 Mar 1;22(3):725-732. doi: 10.31557/APJCP.2021.22.3.725. PMID 33773535
- [Background] Rock CL, Thomson CA, Sullivan KR, Howe CL, Kushi LH, Caan BJ, Neuhouser ML, Bandera EV, Wang Y, Robien K, Basen-Engquist KM, Brown JC, Courneya KS, Crane TE, Garcia DO, Grant BL, Hamilton KK, Hartman SJ, Kenfield SA, Martinez ME, Meyerhardt JA, Nekhlyudov L, Overholser L, Patel AV, Pinto BM, Platek ME, Rees-Punia E, Spees CK, Gapstur SM, McCullough ML. American Cancer Society nutrition and physical activity guideline for cancer survivors. CA Cancer J Clin. 2022 May;72(3):230-262. doi: 10.3322/caac.21719. Epub 2022 Mar 16. PMID 35294043
- [Background] Chaddock-Heyman L, Mackenzie MJ, Zuniga K, Cooke GE, Awick E, Roberts S, Erickson KI, McAuley E, Kramer AF. Higher cardiorespiratory fitness levels are associated with greater hippocampal volume in breast cancer survivors. Front Hum Neurosci. 2015 Aug 26;9:465. doi: 10.3389/fnhum.2015.00465. eCollection 2015. PMID 26379528
- [Background] Naumann F, Martin E, Philpott M, Smith C, Groff D, Battaglini C. Can counseling add value to an exercise intervention for improving quality of life in breast cancer survivors? A feasibility study. J Support Oncol. 2012 Sep-Oct;10(5):188-94. doi: 10.1016/j.suponc.2011.09.004. Epub 2011 Dec 14. PMID 22169703
- [Background] Morrison KS, Paterson C, Toohey K. The Feasibility of Exercise Interventions Delivered via Telehealth for People Affected by Cancer: A Rapid Review of the Literature. Semin Oncol Nurs. 2020 Dec;36(6):151092. doi: 10.1016/j.soncn.2020.151092. Epub 2020 Nov 20. PMID 33223409
- [Background] Sherman KA, Heard G, Cavanagh KL. Psychological effects and mediators of a group multi-component program for breast cancer survivors. J Behav Med. 2010 Oct;33(5):378-91. doi: 10.1007/s10865-010-9265-9. Epub 2010 May 26. PMID 20502954